CLINICAL TRIAL: NCT03319550
Title: Whey vs Casein to Combat Post-inflammatory Protein and Muscle Waste - Combining Endotoxemia, Immobilisation and Fasting in Healthy Young Males in a New Model of Acute Febrile Disease
Brief Title: Whey vs Casein to Combat Post-inflammatory Protein and Muscle Waste in Acute Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Arla Food for Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: theproteinstudy
Record Dates: First submitted 2017-10-13; First posted 2017-10-24 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2018-11

CONDITIONS: Muscle Protein Synthesis; Endotoxemia; Nutrition; Milk Protein; Metabolism; Whey; Casein
Keywords: milk protein, endotoxemia, muscle protein synthesis, whey, casein
MeSH Terms: conditions — Endotoxemia | interventions — Caseins; Whey

STUDY DESIGN:
Intervention Model Description: Interventions*:
  I. LPS (1 ng/kg as bolus) + 36 h fasting + 36 h bedrest + Casein
  II. LPS (1 ng/kg as bolus) + 36 h fasting + 36 h bedrest + Whey
  III. LPS (1 ng/kg as bolus) + 36 h fasting + 36 h bedrest + Leucine-enriched whey
  * LPS will be administered on study day 1 and measurements of metabolism will be performed on study day 2 where we see the secondary effects of acute inflammation. The patient will stay at the hospital over night to ensure continues fast and bedrest.
  The beverages will be isocaloric and with the same total protein content. The basal period will be 2,5 hour with infusion of tracer. Hereafter a total amount of 0,6 g protein/kg bodyweight will be orally administered, 1/3 as a bolus and 2/3 as sipping over 3,5 hours. Muscle biopsies and blodsampels will be collected during both the basal and the sipping period.
Who Masked: Participant, Investigator
Masking Description: The three different protein supplements will be fabricated with the same taste, colour and weight. They will be named "A", "B" and "C" and the investigator will not know which protein is which until all data has been collected and analysed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Casein (Experimental): "LPS + 36 hour fast and bedrest" + Casein (9% leucine) - 0.6 g protein/kg bodyweight, 1/3 as bolus and 2/3 as sipping.
  Interventions: Dietary Supplement: Casein
- Whey (Experimental): "LPS + 36 hour fast and bedrest" + Whey (11% leucine) - 0.6 g protein/kg bodyweight, 1/3 as bolus and 2/3 as sipping
  Interventions: Dietary Supplement: Whey
- Leucine-enriched whey (Experimental): "LPS + 36 hour fast and bedrest" + Leucine-enriched whey (16% leucine) - 0.6 g protein/kg bodyweight, 1/3 as bolus and 2/3 as sipping
  Interventions: Dietary Supplement: Leucine-enriched whey

INTERVENTIONS:
Dietary Supplement: Casein — see experimental description
  Arms: Casein
Dietary Supplement: Whey — see experimental description
  Arms: Whey
Dietary Supplement: Leucine-enriched whey — see experimental description
  Arms: Leucine-enriched whey

SUMMARY:
This study compares three different protein supplements (casein, whey and leucine-enriched whey) and their effect on post-inflammatory muscle waste in a model of acute disease. Each test person will undergo all three interventions.

It is believed that leucine is the primary driver of muscle protein synthesis and therefore we hypothesize that leucine-enriched whey and whey are superior to casein in combating post-inflammatory muscle waste, because of its higher leucine content (16%, 11% and 9% leucine, respectively).

DETAILED DESCRIPTION:
Background:

Acute illness is accompanied by infection/inflammation, anorexia and immobilization all contributing to muscle loss, making nutritional supplement optimization an obvious target for investigation and eventually clinical intervention. In the clinical setting large heterogenicity among patients complicates investigations of muscle metabolism during acute illness. Therefore we introduce a disease model by combining "Inflammation + 36 hour fast and bedrest". Inflammation/febrile illness will be initiated by using the well-established "human endotoxemia model" with a bolus injection of Escherichia coli lipopolysaccharide (LPS), known to cause inflammation comparable with the initial phase of sepsis. The amino acid leucine has shown to be particularly anabolic in performance sports, but little is known about its potential beneficial effects during acute illness. Leucine is a powerful activator of muscle protein synthesis and it seems that protein supplements with the highest leucine content elicit a greater increase in protein synthesis than those with a smaller fraction of leucine.

The protein supplements used most in hospitals contain casein derived protein, which has a much lower leucine content than the whey protein compounds typically used in performance sports.

This study compares three different protein supplements.The study is an open, randomized crossover trial. Laboratory technicians, test subjects and investigators will be blinded.

Interventions:

I. LPS (1 ng/kg as bolus) + 36 h fasting + 36 h bedrest + Casein (9% leucine) II. LPS (1 ng/kg as bolus) + 36 h fasting + 36 h bedrest + Whey (11% leucine) III. LPS (1 ng/kg as bolus) + 36 h fasting + 36 h bedrest + Leucine-enriched whey (16% leucine)

The test objects will be given 0,6 g protein/kg, 1/3 as a bolus and 2/3 as sipping over a period of 3,5 hour. Muscle metabolism will be investigated by phenylalanine tracer using the forearm model and total protein metabolism using a carbamide tracer. Through muscle biopsies intracellular signalling pathways will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male
* Age between 20-40
* BMI between 20-30
* Normal health examination and blood samples
* Written informed consent

Exclusion Criteria:

* Immobilisation of an extremity, unless a doctor has declared it fully rehabilitated.
* Allergy against lidocain or latex.
* The use of anabolic steroids
* Disease like: Diabetes, epilepsia, infection, cardiovascular disease.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
Change in muscle phenylalanine netbalance over the forearm muscle | Change from baseline to 3.5 hours after intervention
  Changes of muscle phenylalanine net balance (= arterio(phe conc)-venous(phe conc) x flow) from baseline to 3.5 hours after intervention using the forearm model

SECONDARY OUTCOMES:
Change in whole body protein metabolism measured by a combination of phenylalanine- and tyrosine tracer | Change from baseline to 3.5 hours after intervention
  Changes in whole body protein synthesis rates (umol/kg/h), breakdown rates (umol/kg/h), phenylalanine to tyrosine conversion rates (umol/kg/h) and net balance (umol/kg/h)
Blood enrichment of essential amino acids | At baseline and every 30 minutes during the intervention period (3.5 hours)
  measures of essential amino acids in the blood
Changes in insulin concentrations | At baseline and every 30 minutes during the intervention period (3.5 hours)
  Measures of insulin concentration in blood
Change in Intracellular signalling in muscle measured by western blotting. | Change from baseline and after 2 hours of intervention
  Investigating intracellular activity of muscle metabolism pathways by western blotting.
Energy expenditure | At baseline and after 2.5 hours of intervention
  Using indirect calorimetry for 15 min
Changes in Glucose, fat and protein oxidation rates | At baseline and after 2.5 hours of intervention
  Using indirect calorimetry for 15 min for measuring glucose- (mg/kg/min), fat- (mg/kg/min) and protein oxidation (mg/kg/min)
Change in muscle breakdown and synthesis rates measured by phenylalanine tracer | Change from baseline to 3.5 hours after intervention
  changes from baseline to 3.5 hours after intervention in Ra(phe)=breakdown (umol/kg/h) and Rd(phe)=synthesis rate (umol/kg/h)
Changes in Glucagon concentrations | Change from baseline and to 1 hour and 3.5 hour after the intervention
  Glucagon concentrations in blood
Changes in GIP concentrations | Change from baseline and to 1 hour and 3.5 hour after the intervention
  GIP concentrations in blood
Changes in GLP-1 concentrations | Change from baseline and to 1 hour and 3.5 hour after the intervention
  GLP-1 concentrations in blood
Changes in Glucose concentrations | At baseline and every 30 minutes during the intervention period (3.5 hours)
  Glucose concentrations in blood
Changes in heart rate profile upon repeated LPS exposure | Measured at baseline and 1,2,3,4,5,6 and 24 hours after LPS (6-8 weeks between visit 1,2 and 3)
  heart rate (beats/min)
Changes in temperature profile upon repeated LPS exposure | Measured at baseline and 1,2,3,4,5,6 and 24 hours after LPS (6-8 weeks between visit 1,2 and 3)
  Axillary temperature (celcius)
Changes in blood pressure profile upon repeated LPS exposure | Measured at baseline and 1,2,3,4,5,6 and 24 hours after LPS (6-8 weeks between visit 1,2 and 3)
  blood pressure (mmHg)
Changes in symptom score profile upon repeated LPS exposure | Measured at baseline and 1,2,3,4,5,6 and 24 hours after LPS (6-8 weeks between visit 1,2 and 3)
  symptom score (from 0-5) for nausea, back pain, muscle pain, headache and chills. 0=no symptoms, 5=severe symptoms.
Changes in TNfalfa profile upon repeated LPS exposure | Measured at baseline and 1, 2, 4, 6 and 24 hours after LPS (6-8 weeks between visit 1,2 and 3)
  TNfalfa blood concentrations
Changes in IL-1 profile upon repeated LPS exposure | Measured at baseline and 1, 2, 4, 6 and 24 hours after LPS (6-8 weeks between visit 1,2 and 3)
  IL-1 blood concentrations
Changes in IL-6 profile upon repeated LPS exposure | Measured at baseline and 1, 2, 4, 6 and 24 hours after LPS (6-8 weeks between visit 1,2 and 3)
  IL-6 blood concentrations
Changes in IL-10 profile upon repeated LPS exposure | Measured at baseline and 1, 2, 4, 6 and 24 hours after LPS (6-8 weeks between visit 1,2 and 3)
  IL-10 blood concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Niels Moeller, Professor, Principal Investigator — Institute for clinical Medicine
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
We will analyse all data ourselves

REFERENCES:
- [Derived] Mose M, Moller N, Jessen N, Mikkelsen UR, Christensen B, Rakvaag E, Hartmann B, Holst JJ, Jorgensen JOL, Rittig N. beta-Lactoglobulin Is Insulinotropic Compared with Casein and Whey Protein Ingestion during Catabolic Conditions in Men in a Double-Blinded Randomized Crossover Trial. J Nutr. 2021 Jun 1;151(6):1462-1472. doi: 10.1093/jn/nxab010. PMID 33693737